CLINICAL TRIAL: NCT03748303
Title: Allopregnanolone Regenerative Therapeutic for Early Alzheimer's Disease: IV to IM Bridging Study
Brief Title: Allopregnanolone Regenerative Therapeutic for Early Alzheimer's Disease: Intramuscular Study
Acronym: Allo-IM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Arizona (Other)
Collaborators: University of Southern California (Other); Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Roberta Brinton, Professor, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlloPhase1-IM
Record Dates: First submitted 2018-10-12; First posted 2018-11-20 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer Dementia
Keywords: Alzheimer's disease; Mild cognitive impairment; Dementia; Regenerative therapeutic; Drug development
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia | interventions — Pregnanolone

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Allo IM cohort (Experimental): Allopregnanolone 4-18mg IM, weekly, for 12 weeks.
  Interventions: Drug: Allopregnanolone

INTERVENTIONS:
Drug: Allopregnanolone — Administration of weekly IM injections of Allopregnanolone.
  Other Names: Allo

SUMMARY:
The purpose of this study is to identifying the intramuscular dose equivalent to the 4mg intravenous dose and assess its safety and tolerability as a weekly injection.

DETAILED DESCRIPTION:
The purpose of this bridging study is to advance the therapeutic development of Allopregnanolone (Allo) by using the intramuscular (IM) route of administration as an alternative to the intravenous (IV) route. In order to identify the equivalent IM dose we will conduct pharmacokinetic (PK) analysis previously informed by simulations and modeling. We will recruit a total of 12 participants, both males and females equally distributed, into this single-arm, open-label study.

PK analysis and dose finding will take place for the initial 4 weeks; some participants may not require all 4 weeks of initial dosing to establish maintenance dose. Once maintenance dose is established all participants will receive weekly administration of Allo IM until they complete 12 weeks total of Allo exposure (5 or 6 clinic visits and 6 or 7 home-nurse visits).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Men or postmenopausal women, aged 55 years or older
* Diagnosis of MCI due to AD or mild AD
* In good general health as evidenced by medical history and with no medical contraindications to participation
* MMSE > 20 at screen
* Caregiver willing and capable to accompany the patient to clinic visits

Exclusion Criteria:

* Daily use of benzodiazepines, sedative/hypnotics, anticonvulsants, antipsychotics, and other drugs that might interact with the GABA-A receptor complex.
* Seizure disorder, history of stroke, focal brain lesion, traumatic brain injury, substance abuse, malignancy.
* Clinically significant laboratory or ECG abnormality obtained at screening visit.
* MRI indicative of significant abnormality, including but not limited to evidence of a single prior hemorrhage or infarct >1 cm3, multiple lacunar infarcts (>1) or evidence of a single prior infarct >1cm3, evidence of a cerebral contusion, encephalomalacia, aneurysms, vascular malformations, subdural hematoma, or space occupying lesions (e.g. abscess or tumor).
* Has any contraindications for MRI studies, including claustrophobia, the presence of metal (ferromagnetic) implants, or a cardiac pacemaker that is not compatible with MRI.
* Is currently enrolled in a clinical trial involving an off-label use of an investigational drug or device, or concurrently enrolled in any other type of medical research or observational study judged not to be scientifically or medically compatible with this study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse events | From baseline to visit 16 (14 weeks)
  Incidence and severity of treatment emergent adverse events assessed weekly.
Safety - clinical laboratory measures | From Baseline to visit 16 (14 weeks)
  Proportion of subjects exceeding pre-established critical laboratory values.
Safety - clinical assessment | From Baseline to visit 16 (14 weeks)
  Proportion of subjects with abnormal findings in physical/neurological exams, vital signs and electrocardiograms.

SECONDARY OUTCOMES:
Pharmacokinetic parameter - Cmax | Visits 3 - 6 (up to 4 weeks)
  Determine maximum serum concentration of Allo after IM administration of each dose.
Pharmacokinetic parameter - AUC | Visits 3 - 6 (up to 4 weeks)
  Determine the area under the curve after each IM administration of Allo.
Pharmacokinetic parameter - Tmax | Visits 3 - 6 (up to 4 weeks)
  Determine the time at which Cmax is attained.
Pharmacokinetic parameter - Clearance | Visits 3 - 6 (up to 4 weeks)
  Pharmacokinetic measurement of the volume of plasma from which Allo is completely removed per unit time.
Pharmacokinetic parameter - Volume of distribution | Visits 3 - 6 (up to 4 weeks)
  Determine the volume of distribution at steady state of Allo.
Satisfaction and feasibility of home nurse survey | Visits 8-9 and 11-15 (up to 8 weeks)
  Standardized patient satisfaction questionnaire to assess the feasibility of home-health care visits to administer the study medication and its desirability by participants and caregivers. Levels of satisfaction measured on a 5-point scale (1 = lowest satisfaction, 5 = greatest).

OTHER OUTCOMES:
MRI brain volumes | Baseline to visit 16 (14 weeks)
  To evaluate MRI-based brain volumes 1-week before before and 1-week after the administration of Allo IM for 12 weeks (total assessment period of 14 weeks).
Cambridge Neuropsychological Test Automated Battery (CANTAB) Paired Associates Learning (PAL) | Baseline to visit 16 (14 weeks)
  Test to evaluate changes in cognition
Mini-Mental State Exam (MMSE) | Baseline to visit 16 (14 weeks)
  Test to evaluate changes in cognition.
Alzheimer's Disease Assessment Scale Cognitive Subscale 14 (ADAS-Cog14) | Baseline to visit 16 (14 weeks)
  Well known test to evaluate changes in cognition. Scores on this 14 item test range from 0 (best) to 85 (worse); a positive change indicates cognitive worsening.
Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) | Baseline to visit 16 (14 weeks)
  Clinical scale that rates the severity of dementia as absent, questionable, mild, moderate, or severe (CDR score of 0, 0.5, 1, 2, or 3, respectively).
Cogstate Alzheimer's battery | Baseline to visit 16 (14 weeks)
  Test to evaluate changes in cognition.
Activities of daily living | Baseline to visit 16 (14 weeks)
  To assess activities of daily living per the Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale (ADCS-iADLS). In a structured interview format, informants are queried as to whether participants attempted each item in the inventory during the prior 4 weeks and their level of performance. Scores range from 0-56.
Caregiver burden survey | Baseline to visit 16 (14 weeks)
  Assessed per Zarit's burden 22-item questionnaire. Burden measured on a 5-point scale (0 = never burdened, 4 = nearly always burdened). Max score = 88
Actigraphy sleep assessment - Total sleep time | Screen to visit 16 (16 weeks)
  To assess standard sleep parameters using wearable devices (actigraph wristwatch): Total sleep time reported as time in minutes.
Actigraphy sleep assessment - Wake after sleep onset | Screen to visit 16 (16 weeks)
  To assess standard sleep parameters using wearable devices (actigraph wristwatch): Wake after sleep onset (WASO) reported as time in minutes.
Actigraphy sleep assessment - Sleep efficiency | Screen to visit 16 (16 weeks)
  To assess standard sleep parameters using wearable devices (actigraph wristwatch): Sleep efficiency reported as percentage.
Physical activity | Screen to visit 16 (16 weeks)
  To assess daily activity using wearable devices: FitBit.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta D Brinton, PhD, Principal Investigator — University of Arizona; Lon S Schneider, MD, MS, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California - Alzheimer Disease Research Center - Healthcare Consultation Center II, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided